CLINICAL TRIAL: NCT01639430
Title: Diagnostic Accuracy of Body Temperature Measurement in Geriatric Patients Presenting to the Emergency Department
Brief Title: Diagnostic Accuracy of Body Temperature Measurement in Geriatric Patients
Status: Completed | Type: Observational
Sponsor: Klinikum Nürnberg (Other)
Responsible Party: Principal Investigator, Dr. Katrin Singler, senior physician, Klinikum Nürnberg
Other Study IDs: KSMC-tempger-1
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Fever; Infection
MeSH Terms: conditions — Fever; Infections | interventions — Administration, Rectal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Geriatric patients ED: Consecutive patients >= 75 years in the emergency department.
  Interventions: Other: rectal, tympanal and temporal artery thermometry

INTERVENTIONS:
Other: rectal, tympanal and temporal artery thermometry — Temperature measurement was done once in all patients included within the first hour of patients´presentation to the emergency department.
  Tympanal measurement was carried out by the use of infrared ear thermometry, temporal artery thermometry was done using infrared technology as well.

SUMMARY:
Retrospective analysis of a quality measurement project examining the quality of vital parameter measurement in consecutive patients >= 75 years presenting to the emergency department.

Primary goal of the study is to evaluate the diagnostic accuracy of body temperature measurement using different methods to diagnose infection in patients >= 75 years presenting to the emergency department. The secondary goal is to compare the reliability of tympanal and temporal artery thermometry with rectal temperature measurement.

ELIGIBILITY:
Inclusion Criteria:

* >= 75 years
* given informed consent

Exclusion Criteria:

* patients who do not speak the German language
* patients with unstable cardiorespiratory status
* presence of contraindications to one of the temperature measurement methods

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Consecutive patients >= 75 years presenting to the emergency department of an urban university-affiliated hospital (80.000 attendees per year).
Sampling Method: Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of rectal, tympanal and temporal artery thermometry to diagnose infection | June 2012
  The primary outcome measure is the diagnostic accuracy of rectal, tympanal and temporal artery thermometry to diagnose infection in old patients presenting to the ED

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Nürnberg, emergency department, Nuremberg, Bavaria, Germany